CLINICAL TRIAL: NCT02369965
Title: Efficacy and Safety of Albuvirtide for Injection Combined With LPV/r for Treatment of HIV-1-Infected Patients Failed First-line Antiretroviral Therapy
Brief Title: Test Albuvirtide in Experienced Patients
Acronym: TALENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FB-ABWT-Ⅲ-301; ChiCTR-TRC-14004276 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: HIV Infections; AIDS
Keywords: HIV-1; AIDS; Albuvirtide; Treatment-experienced; Fusion inhibitor
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — albuvirtide; Lopinavir; lopinavir-ritonavir drug combination; Tenofovir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albuvirtide, lopinavir-ritonavir (Experimental): albuvirtide once a week and lopinavir-ritonavir twice daily for 48 weeks
  Interventions: Drug: albuvirtide; Drug: lopinavir-ritonavir
- lopinavir-ritonavir,tenofovir,lamivudine (Active Comparator): lopinavir-ritonavir twice daily, tenofovir once daily and lamivudine once daily for 48 weeks
  Interventions: Drug: lopinavir-ritonavir; Drug: tenofovir; Drug: lamivudine

INTERVENTIONS:
Drug: albuvirtide — albuvirtide 320mg administered intravenously once a week
  Other Names: ABT
  Arms: albuvirtide, lopinavir-ritonavir
Drug: lopinavir-ritonavir — lopinavir-ritonavir 400/100mg administered orally twice daily
  Other Names: Kaletra; LPV/r
Drug: tenofovir — tenofovir 300mg administered orally once daily
  Other Names: TDF
  Arms: lopinavir-ritonavir,tenofovir,lamivudine
Drug: lamivudine — lamivudine 300mg administered orally once daily
  Other Names: 3TC
  Arms: lopinavir-ritonavir,tenofovir,lamivudine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of albuvirtide combined with lopinavir-ritonavir (LPV/r) in HIV-1-infected patients who failed first-line antiretroviral therapy (ART).

DETAILED DESCRIPTION:
This was a 48-week, multi-center, open-label, randomized and controlled, non-inferiority phase 3 clinical trial to evaluate the safety and efficacy of albuvirtide combined with LPV/r in HIV-1 infected patients who failed their first-line ART and had HIV-1 RNA levels ≥ 1000 copies/mL at screening.

The trial was conducted in 12 sites in China. Subjects meeting inclusion criteria were randomized in a 1:1 ratio to ABT group and NRTI group, in which the ABT group received albuvirtide and LPV/r combination therapy, and NRTI group received the standard 3-drug regimen of LPV/r + Lamivudine (3TC) + Tenofovir (TDF). If TDF was used in the previous regimen or genotypic resistance histories showed primary mutation to TDF, zidovudine (AZT) or abacavir (ABC) would be used. Albuvirtide was given by weekly intravenous infusion and LPV/r was given twice daily orally. A total of 418 subjects were randomized, of whom 401 received at least one treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 16-60 years old, male or female.
2. Those who meet the Diagnostic Criteria of AIDS and HIV Infection, the Health Industry Standard of the People's Republic of China (WS 293-2008).
3. Those who have been undergoing antiretroviral treatment with nucleosides and non-nucleoside reverse transcriptase inhibitors (NRTIs+NNRTIs) for at least 6 months.
4. HIV-RNA ≥ 1000 copies/mL.
5. Those who have no serious hepatic or renal functional impairment and other parameters are generally in the normal ranges according to the comprehensive physical examinations (including general physical examination, routine blood and urine tests, blood chemistry tests, ECG, etc.).
6. The subjects should have a full understanding of the objective, nature, methods of the trial and the possible reactions. He/She should participate in the trial voluntarily and should sign the informed consent form.

Exclusion Criteria:

1. Those who are in an acute stage of infection, or have suffered from AIDS-related diseases (e.g. opportunistic infections or malignant tumors, etc.) at enrollment; or have suffered from opportunistic infections within 3 months prior to enrollment and the conditions have not reached a stable state within 2 weeks prior to enrollment.
2. Those who have used protease inhibitors or HIV fusion inhibitors for antiretroviral treatment, and who have participated in HIV vaccine clinical trials or have participated in other drug trials within recent 3 months.
3. Those who have been co-administered antiviral treatment for hepatitis.
4. Those whose screening test results meet one of the following: hemoglobin < 9 g/dL, WBC count <2×109/L, neutrophil count < 1×109/L, PLT count < 75×109/L, transaminase > 3×ULN, total bilirubin > 2×ULN, creatinine > 1×ULN, serum creatine phosphokinase > 2×ULN.
5. Those with allergic constitution or known allergic to ingredients of the investigational drug or ART drugs prescribed in the protocol.
6. Currently suffering from serious chronic diseases, metabolic diseases (such as diabetes mellitus), neurological and psychiatric disorders.
7. Patients with hemophilia A or B.
8. Those with suspected or confirmed history of alcohol or drug abuse.
9. Pregnant or lactating women; or women of childbearing age who refuse to take contraceptive measures during the trial.
10. Those for whom the possibility of being enrolled is low according to the judgment of the investigator (e.g. weak physical condition, poor compliance, etc.).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 418 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants of virological suppression at Week 48 | Through Week 48
  Percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48

SECONDARY OUTCOMES:
Changes of viral load | Baseline to Week 48
  Changes of HIV-1 RNA relative to baseline at Week 48
Percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48 | Through Week 48
  Percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48
Changes of CD4 cell count | Baseline to Week 48
  Changes of CD4 cell count relative to baseline at Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Dong Xie, Study Director — Frontier Biotechnologies Inc.
Locations (12):
- China (12):
  - 302 Hospital People's Liberation Army Of China, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital medical university, Beijing, Beijing Municipality
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - The Third People'S Hospital Of Shenzhen, Shenzhen, Guangdong
  - Henan Infectious Disease Hospital, Zhengzhou, Henan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - Affiliated Hangzhou Xixi Hospital,Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Su B, Yao C, Zhao QX, Cai WP, Wang M, Lu HZ, Chen YY, Liu L, Wang H, He Y, Zheng YH, Li LH, Chen JF, Yu JH, Zhu B, Zhao M, Sun YT, Lun WH, Xia W, Sun LJ, Dai LL, Jiang TY, Wang MX, Zheng QS, Peng HY, Wang Y, Lu RJ, Hu JH, Xing H, Shao YM, Xie D, Zhang T, Zhang FJ, Wu H; TALENT Study Team. Efficacy and safety of the long-acting fusion inhibitor albuvirtide in antiretroviral-experienced adults with human immunodeficiency virus-1: interim analysis of the randomized, controlled, phase 3, non-inferiority TALENT study. Chin Med J (Engl). 2020 Nov 25;133(24):2919-2927. doi: 10.1097/CM9.0000000000001273. PMID 33252379